CLINICAL TRIAL: NCT04936035
Title: A Randomized, Double-blind, Placebo-Controlled, Dose-Ranging Multicenter Study to Evaluate the Efficacy and Safety of ALN-AGT01 in Patients With Mild-to-Moderate Hypertension
Brief Title: A Study to Evaluate Efficacy and Safety of ALN-AGT01 in Patients With Mild To-Moderate Hypertension
Acronym: KARDIA-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALN-AGT01-002; 2021-001248-82 (EudraCT Number)
Record Dates: First submitted 2021-06-14; First posted 2021-06-23 (Actual); Results first posted 2024-12-27 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Hypertension
Keywords: High blood pressure; Hypertension; Hypertensive; siRNA; Angiotensinogen; AGT
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Placebo (Placebo Comparator): Participants received zilebesiran matching placebo, subcutaneous (SC) injection, once every 3 months (Q3M), with re-randomization at Month 6 to 1 of the initial 4 zilebesiran regimens. Participants will continue their respective zilebesiran regimen up to Month 12 in the DB period and up to 24 additional months in the DB Extension period. Upon implementation of Amendment 6, the DB Extension period was closed.
  Interventions: Drug: Placebo; Drug: ALN-AGT01
- Zilebesiran 150 Milligrams (mg) Once Every 6 Months (Q6M) (Experimental): Participants receive zilebesiran, 150 mg, SC injection, Q6M, during the 12-month DB period. Participants will continue receiving the same zilebesiran regimen for up to 24 additional months in the DB Extension period. Participants in this arm will receive a placebo during those dosing visits when they do not receive zilebesiran to maintain the blind. Upon implementation of Amendment 6, the DB Extension period was closed.
  Interventions: Drug: Placebo; Drug: ALN-AGT01
- Zilebesiran 300 mg Q6M (Experimental): Participants receive zilebesiran, 300 mg, SC injection, Q6M, during the 12-month DB period. Participants will continue receiving the same zilebesiran regimen for up to 24 additional months in the DB Extension period. Participants in this arm will receive a placebo during those dosing visits when they do not receive zilebesiran to maintain the blind. Upon implementation of Amendment 6, the DB Extension period was closed.
  Interventions: Drug: Placebo; Drug: ALN-AGT01
- Zilebesiran 300 mg Q3M (Experimental): Participants receive zilebesiran, 300 mg, SC injection, Q3M, during the 12-month DB period. Participants continue receiving the same zilebesiran regimen for up to 24 additional months in the DB Extension period. Upon implementation of Amendment 6, the DB Extension period was closed.
  Interventions: Drug: ALN-AGT01
- Zilebesiran 600 mg Q6M (Experimental): Participants receive zilebesiran, 600 mg, SC injection, Q6M, during the 12-month DB period. Participants will continue receiving the same zilebesiran regimen for up to 24 additional months in the DB Extension period. Participants in this arm will receive a placebo during those dosing visits when they do not receive zilebesiran to maintain the blind. Upon implementation of Amendment 6, the DB Extension period was closed.
  Interventions: Drug: Placebo; Drug: ALN-AGT01

INTERVENTIONS:
Drug: Placebo — Placebo administered by SC injection
  Arms: Placebo; Zilebesiran 150 Milligrams (mg) Once Every 6 Months (Q6M); Zilebesiran 300 mg Q6M; Zilebesiran 600 mg Q6M
Drug: ALN-AGT01 — ALN-AGT01 administered by SC injection
  Other Names: Zilebesiran

SUMMARY:
The purpose of this study is to evaluate the effect of ALN-AGT01 on systolic and diastolic blood pressure and to characterize the pharmacodynamic (PD) effects and safety of ALN-AGT01.

DETAILED DESCRIPTION:
Participants will receive ALN-AGT01 or placebo for the first 6 months of the 12-month double-blind (DB) treatment period. Participants randomized to placebo will be re-randomized at Month 6 to 1 of the 4 initial ALN-AGT01 regimens until the end of the 12-month DB treatment period. Participants randomized to ALN-AGT01 regimens will remain on their originally assigned regimens through remainder of the study.

ELIGIBILITY:
Inclusion Criteria:

* Daytime mean SBP ≥135 mmHg and ≤160 mmHg by ABPM, without antihypertensive medication

Exclusion Criteria:

* Secondary hypertension, orthostatic hypotension
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2× upper limit of normal (ULN)
* Elevated potassium >5 mEq/L
* Estimated glomerular filtration rate (eGFR) of ≤30 mL/min/1.73m^2
* Received an investigational agent within the last 30 days
* Type 1 diabetes mellitus, poorly controlled Type 2 diabetes mellitus, newly diagnosed Type 2 diabetes mellitus
* History of any cardiovascular event within 6 months prior to randomization
* History of intolerance to SC injection(s)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 394 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2024-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Alnylam Pharmaceuticals
Locations (68):
- United States (47):
  - Clinical Trial Site, Birmingham, Alabama
  - Clinical Trial Site, Tempe, Arizona
  - Clinical Trial Site, Beverly Hills, California
  - Clinical Trial Site, La Mesa, California
  - Clinical Trial Site, Los Angeles, California
  - Clinical Trial Site, San Diego, California
  - Clinical Trial Site, South Gate, California
  - Clinical Trial Site, Vista, California
  - Clinical Trial Site, Washington D.C., District of Columbia
  - Clinical Trial Site, Clearwater, Florida
  - Clinical Trial Site, Coral Gables, Florida
  - Clinical Trial Site, Fleming Island, Florida
  - Clinical Trial Site, Hollywood, Florida
  - Clinical Trial Site, Inverness, Florida
  - Clinical Trial Site, Jacksonville, Florida
  - Clinical Trial Site, Miami, Florida
  - Clinical Trial Site, Naples, Florida
  - Clinical Trial Site, Orlando, Florida
  - Clinical Trial Site, Acworth, Georgia
  - Clinical Trial Site, Columbus, Georgia
  - Clinical Trial Site, Fayetteville, Georgia
  - Clinical Trial Site, Macon, Georgia
  - Clinical Trial Site, Champaign, Illinois
  - Clinical Trial Site, Valparaiso, Indiana
  - Clinical Trial Site, West Des Moines, Iowa
  - Clinical Trial Site, Lake Charles, Louisiana
  - Clinical Trial Site, New Orleans, Louisiana
  - Clinical Trial Site, Prairieville, Louisiana
  - Clinical Trial Site, Baltimore, Maryland
  - Clinical Trial Site, Jackson, Mississippi
  - Clinical Trial Site, Jefferson City, Missouri
  - Clinical Trial Site, Las Vegas, Nevada
  - Clinical Trial Site, New York, New York
  - Clinical Trial Site, The Bronx, New York
  - Clinical Trial Site, Greensboro, North Carolina
  - Clinical Trial Site, Medford, Oregon
  - Clinical Trial Site, Greenville, South Carolina
  - Clinical Trial Site, Memphis, Tennessee
  - Clinical Trial Site, Cedar Park, Texas
  - Clinical Trial Site, Houston, Texas
  - Clinical Trial Site, Magnolia, Texas
  - Clinical Trial Site, Pearland, Texas
  - Clinical Trial Site, San Antonio, Texas
  - Clinical Trial Site, Stephenville, Texas
  - Clinical Trial Site, Tomball, Texas
  - Clinical Trial Site, Waco, Texas
  - Clinical Trial Site, Burke, Virginia
- Canada (10):
  - Clinical Trial Site, Red Deer, Alberta
  - Clinical Trial Site, New Minas, Nova Scotia
  - Clinical Trial Site, Brampton, Ontario
  - Clinical Trial Site, Toronto, Ontario
  - Clinical Trial Site, Chicoutimi, Quebec
  - Clinical Trial Site, Mirabel, Quebec
  - Clinical Trial Site, Montreal, Quebec
  - Clinical Trial Site, Québec, Quebec
  - Clinical Trial Site, Trois-Rivières, Quebec
  - Clinical Trial Site, Victoriaville, Quebec
- Puerto Rico (3):
  - Clinical Trial Site, Bayamón
  - Clinical Trial Site, Ponce
  - Clinical Trial Site, San Juan
- Ukraine (4):
  - Clinical Trial Site, Ivano-Frankivsk
  - Clinical Trial Site, Kharkiv
  - Clinical Trial Site, Odesa
  - Clinical Trial Site, Uzhhorod
- United Kingdom (4):
  - Clinical Trial Site, Glasgow
  - Clinical Trial Site, Hexham
  - Clinical Trial Site, London
  - Clinical Trial Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Access to Anonymized individual participant data that support these results is made available 12 months after study completion and not less than 12 months after the product and indication have been approved in the US and/or the EU.
  Data will be provided contingent upon the approval of a research proposal and the execution of a data sharing agreement. Requests for access to data can be submitted via the website www.vivli.org.

REFERENCES:
- [Derived] Bakris GL, Saxena M, Gupta A, Chalhoub F, Lee J, Stiglitz D, Makarova N, Goyal N, Guo W, Zappe D, Desai AS; KARDIA-1 Study Group. RNA Interference With Zilebesiran for Mild to Moderate Hypertension: The KARDIA-1 Randomized Clinical Trial. JAMA. 2024 Mar 5;331(9):740-749. doi: 10.1001/jama.2024.0728. PMID 38363577

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total of 86 clinical sites across North America & 25 sites in Europe enrolled 394 participants. 16 participants from Ukraine were unable to continue participation due to geopolitical instability. Due to challenges in data collection & cleaning, these participants were excluded from all analysis sets. Hence, results are presented for 378 randomized participants. Study has 2 periods: 6-Month Placebo-controlled Double-blind (DB) Period & Post-6-Month DB Period [DB (Months 6 to 12)+DB Extension].
Pre-assignment Details: As pre-specified in SAP, data collected for the participant flow after '6-Month Placebo-controlled DB Period' (i.e., Months 6 to 12 DB period + DB Extension Period) was to be reported together as 'Post-6-Month DB Period' per treatment sequence (Pbo/Zil & Zil/Zil). Before Protocol Amendment 6 (PA6), participants completing 12 months in this study could join a separate open-label extension (OLE) study. With PA6, the OLE study was canceled. Hence, the 24-month extension treatment was also ended.
Groups:
- Placebo: Participants received zilebesiran matching placebo, as subcutaneous (SC) injection, once every 3 months (Q3M) during the 6-month placebo-controlled double-blind (DB) period.
- Zilebesiran 150 Milligrams (mg) Once Every 6 Months (Q6M): Participants received zilebesiran, 150 mg, as SC injection on Day 1 of the 6-month placebo-controlled DB period. They received placebo at Month 3 of the 6-month placebo-controlled DB period to maintain the blind.
- Zilebesiran 300 mg Q6M: Participants received zilebesiran, 300 mg, as SC injection on Day 1 of the 6-month placebo-controlled DB period. They received placebo at Month 3 of the 6-month placebo-controlled DB period to maintain the blind.
- Zilebesiran 300 mg Q3M: Participants received zilebesiran, 300 mg, as SC injection, Q3M, during the 6-month placebo-controlled DB period.
- Zilebesiran 600 mg Q6M: Participants received zilebesiran, 600 mg, as SC injection, on Day 1 of the 6-month placebo-controlled DB period. They received placebo at Month 3 of the 6-month placebo-controlled DB period to maintain the blind.
- Placebo/Zilebesiran 150 mg Q6M: Participants who received placebo during the 6-month placebo-controlled DB period were re-randomized at Month 6 to 1 of the 4 initial zilebesiran regimens. Participants in this arm received zilebesiran, 150 mg, as SC injection Q6M after re-randomization for the remainder of the study. Participants received placebo at the visit where no zilebesiran dose was planned to maintain blind between the Q3M and Q6M regimens.
  Prior to PA6, participants who completed Months 6 to 12 of blinded treatment and pre-dose assessment at Month 12, before a separate OLE study was available, could continue receiving blinded zilebesiran treatment up to additional 24 months in the DB Extension Period. Following PA6, the DB Extension Period was discontinued. Participants who had not yet completed the Month 12 visit at the time of PA6 implementation received their last dose of study drug at Month 9. For participants already in the DB Extension Period at the time of PA6 implementation, dosing depended on scheduled visits: participants whose next visit was at Month 15, 21, 27, or 33 received their planned study drug, while those whose next visit was at Month 18, 24, 30, or 36 did not receive further study drug in the study.
- Placebo/Zilebesiran 300 mg Q6M: Participants who received placebo during the 6-month placebo-controlled DB period were re-randomized at Month 6 to 1 of the 4 initial zilebesiran regimens. Participants in this arm received zilebesiran, 300 mg, as SC injection Q6M after re-randomization for the remainder of the study. Participants received placebo at the visit where no zilebesiran dose was planned to maintain blinding between the Q3M and Q6M regimens.
  Prior to PA6, participants who completed Months 6 to 12 of blinded treatment and pre-dose assessment at Month 12, before a separate OLE study was available, could continue receiving blinded zilebesiran treatment up to additional 24 months in the DB Extension Period. Following PA6, the DB Extension Period was discontinued. Participants who had not yet completed the Month 12 visit at the time of PA6 implementation received their last dose of study drug at Month 9. For participants already in the DB Extension Period at the time of PA6 implementation, dosing depended on scheduled visits: participants whose next visit was at Month 15, 21, 27, or 33 received their planned study drug, while those whose next visit was at Month 18, 24, 30, or 36 did not receive further study drug in the study.
- Placebo/Zilebesiran 300 mg Q3M: Participants who received placebo during 6-month placebo-controlled DB period were re-randomized at Month 6 to 1 of the 4 initial zilebesiran regimens. Participants in this arm received zilebesiran, 300 mg, as SC injection Q3M after re-randomization for the remainder of the study.
  Prior to PA6, participants who completed Months 6 to 12 of blinded treatment and pre-dose assessment at Month 12, before a separate OLE study was available, could continue receiving blinded zilebesiran treatment up to additional 24 months in the DB Extension Period. Following PA6, the DB Extension Period was discontinued. Participants who had not yet completed the Month 12 visit at the time of PA6 implementation received their last dose of study drug at Month 9. For participants already in the DB Extension Period at the time of PA6 implementation, dosing depended on scheduled visits: participants whose next visit was at Month 15, 21, 27, or 33 received their planned study drug, while those whose next visit was at Month 18, 24, 30, or 36 did not receive further study drug in the study.
- Placebo/Zilebesiran 600 mg Q6M: Participants who received placebo 6-month placebo-controlled DB period were re-randomized at Month 6 to 1 of the 4 initial zilebesiran regimens. Participants in this arm received zilebesiran, 600 mg, as SC injection Q6M after re-randomization for the remainder of the study. Participants received placebo at the visit where no zilebesiran dose was planned to maintain blinding between the Q3M and Q6M regimens.
  Prior to PA6, participants who completed Months 6 to 12 of blinded treatment and pre-dose assessment at Month 12, before a separate OLE study was available, could continue receiving blinded zilebesiran treatment up to additional 24 months in the DB Extension Period. Following PA6, the DB Extension Period was discontinued. Participants who had not yet completed the Month 12 visit at the time of PA6 implementation received their last dose of study drug at Month 9. For participants already in the DB Extension Period at the time of PA6 implementation, dosing depended on scheduled visits: participants whose next visit was at Month 15, 21, 27, or 33 received their planned study drug, while those whose next visit was at Month 18, 24, 30, or 36 did not receive further study drug in the study.
- Zilebesiran/Zilebesiran 150 mg Q6M: Participants who received zilebesiran 150 mg Q6M during the 6-month placebo-controlled DB period remained on the same regimen throughout the study. Participants received placebo at the visit where no zilebesiran dose was planned to maintain blinding between the Q3M and Q6M regimens.
  Prior to PA6, participants who completed Months 6 to 12 of blinded treatment and pre-dose assessment at Month 12, before a separate OLE study was available, could continue receiving blinded zilebesiran treatment up to additional 24 months in the DB Extension Period. Following PA6, the DB Extension Period was discontinued. Participants who had not yet completed the Month 12 visit at the time of PA6 implementation received their last dose of study drug at Month 9. For participants already in the DB Extension Period at the time of PA6 implementation, dosing depended on scheduled visits: participants whose next visit was at Month 15, 21, 27, or 33 received their planned study drug, while those whose next visit was at Month 18, 24, 30, or 36 did not receive further study drug in the study.
- Zilebesiran/Zilebesiran 300 mg Q6M: Participants who received zilebesiran 300 mg Q6M during the 6-month placebo-controlled DB period remained on the same regimen throughout the study. Participants received placebo at the visit where no zilebesiran dose was planned to maintain blinding between the Q3M and Q6M regimens.
  Prior to PA6, participants who completed Months 6 to 12 of blinded treatment and pre-dose assessment at Month 12, before a separate OLE study was available, could continue receiving blinded zilebesiran treatment up to additional 24 months in the DB Extension Period. Following PA6, the DB Extension Period was discontinued. Participants who had not yet completed the Month 12 visit at the time of PA6 implementation received their last dose of study drug at Month 9. For participants already in the DB Extension Period at the time of PA6 implementation, dosing depended on scheduled visits: participants whose next visit was at Month 15, 21, 27, or 33 received their planned study drug, while those whose next visit was at Month 18, 24, 30, or 36 did not receive further study drug in the study.
- Zilebesiran/Zilebesiran 300 mg Q3M: Participants who received zilebesiran 300 mg Q3M during the 6-month placebo-controlled DB period remained on the same regimen throughout the study.
  Prior to PA6, participants who completed Months 6 to 12 of blinded treatment and pre-dose assessment at Month 12, before a separate OLE study was available, could continue receiving blinded zilebesiran treatment up to additional 24 months in the DB Extension Period. Following PA6, the DB Extension Period was discontinued. Participants who had not yet completed the Month 12 visit at the time of PA6 implementation received their last dose of study drug at Month 9. For participants already in the DB Extension Period at the time of PA6 implementation, dosing depended on scheduled visits: participants whose next visit was at Month 15, 21, 27, or 33 received their planned study drug, while those whose next visit was at Month 18, 24, 30, or 36 did not receive further study drug in the study.
- Zilebesiran/Zilebesiran 600 mg Q6M: Participants who received zilebesiran 600 mg Q6M during the 6-month placebo-controlled DB period remained on the same regimen throughout the study. Participants received placebo at the visit where no zilebesiran dose was planned to maintain blinding between the Q3M and Q6M regimens.
  Prior to PA6, participants who completed Months 6 to 12 of blinded treatment and pre-dose assessment at Month 12, before a separate OLE study was available, could continue receiving blinded zilebesiran treatment up to additional 24 months in the DB Extension Period. Following PA6, the DB Extension Period was discontinued. Participants who had not yet completed the Month 12 visit at the time of PA6 implementation received their last dose of study drug at Month 9. For participants already in the DB Extension Period at the time of PA6 implementation, dosing depended on scheduled visits: participants whose next visit was at Month 15, 21, 27, or 33 received their planned study drug, while those whose next visit was at Month 18, 24, 30, or 36 did not receive further study drug in the study.
Period: 6-Month Placebo-controlled DB Period
Arm/Group | Placebo | Zilebesiran 150 Milligrams (mg) Once Every 6 Months (Q6M) | Zilebesiran 300 mg Q6M | Zilebesiran 300 mg Q3M | Zilebesiran 600 mg Q6M | Placebo/Zilebesiran 150 mg Q6M | Placebo/Zilebesiran 300 mg Q6M | Placebo/Zilebesiran 300 mg Q3M | Placebo/Zilebesiran 600 mg Q6M | Zilebesiran/Zilebesiran 150 mg Q6M | Zilebesiran/Zilebesiran 300 mg Q6M | Zilebesiran/Zilebesiran 300 mg Q3M | Zilebesiran/Zilebesiran 600 mg Q6M
Started | 76 | 78 | 73 | 75 | 76 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 70 | 70 | 70 | 70 | 71 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 6 | 8 | 3 | 5 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Deviation | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Subject Stopped Participation in the Study | 5 | 5 | 1 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Reason Unknown | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Post-6-Month DB Period (30months)
Arm/Group | Placebo | Zilebesiran 150 Milligrams (mg) Once Every 6 Months (Q6M) | Zilebesiran 300 mg Q6M | Zilebesiran 300 mg Q3M | Zilebesiran 600 mg Q6M | Placebo/Zilebesiran 150 mg Q6M | Placebo/Zilebesiran 300 mg Q6M | Placebo/Zilebesiran 300 mg Q3M | Placebo/Zilebesiran 600 mg Q6M | Zilebesiran/Zilebesiran 150 mg Q6M | Zilebesiran/Zilebesiran 300 mg Q6M | Zilebesiran/Zilebesiran 300 mg Q3M | Zilebesiran/Zilebesiran 600 mg Q6M
Started | 0 | 0 | 0 | 0 | 0 | 17 | 17 | 16 | 18 | 69 | 67 | 66 | 65
Completed Month 12 Visit | 0 | 0 | 0 | 0 | 0 | 13 | 16 | 16 | 18 | 65 | 62 | 65 | 61
Completed | 0 | 0 | 0 | 0 | 0 | 12 | 15 | 15 | 18 | 60 | 57 | 59 | 58
Not Completed | 0 | 0 | 0 | 0 | 0 | 5 | 2 | 1 | 0 | 9 | 10 | 7 | 7
Not completed — Participant Stopped Participation in the Study | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 2 | 7 | 5 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 3 | 1 | 1 | 4
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Reason Not Specified | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set included all randomized participants who received any amount of the study drug.
Groups:
- Placebo: Participants received zilebesiran matching placebo, as SC injection, Q3M during the 6-month placebo-controlled DB period.
- Zilebesiran 150 mg Q6M: Participants received zilebesiran, 150 mg, as SC injection on Day 1 of the 6-month placebo-controlled DB period. They received placebo at Month 3 of the 6-month placebo-controlled DB period to maintain the blind.
- Total: Total of all reporting groups
Arm/Group | Placebo | Zilebesiran 150 mg Q6M | Zilebesiran 300 mg Q6M | Zilebesiran 300 mg Q3M | Zilebesiran 600 mg Q6M | Total
Number analyzed (Participants) | 75 | 78 | 73 | 75 | 76 | 377
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (11.2) | 55.5 (10.6) | 56.4 (10.3) | 57.7 (10.6) | 57.4 (10.2) | 56.8 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 39 | 29 | 30 | 31 | 167
  Male | 37 | 39 | 44 | 45 | 45 | 210
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 19 | 16 | 10 | 20 | 74
  Not Hispanic or Latino | 66 | 59 | 57 | 65 | 56 | 303
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 1
  Asian | 5 | 4 | 2 | 7 | 5 | 23
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 0 | 1
  Black or African American | 18 | 20 | 17 | 19 | 19 | 93
  White | 52 | 53 | 54 | 48 | 52 | 259
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
24-hour Mean Systolic Blood Pressure (SBP) Assessed by Ambulatory Blood Pressure Monitoring (ABPM) [Mean (Standard Deviation); unit: millimeter of mercury (mmHg)] — 24 hour ABPM was programmed to take readings every 20 minutes during day (6 am -9:59 pm) and every 30 minutes during the night (10 pm-5:59 am). ABPM was considered adequate if: 1. the number of successful daytime readings were ≥33, 2. the number of successful nighttime readings were ≥11, 3. no more than 3 hours are not represented (i.e.,3 sections of 60 minutes where 0 valid readings were obtained). To summarize 24 hour ABPM, the hourly adjusted mean was calculated. Hourly mean was the average of blood pressure (BP) by each hour of the day. The 24 hour mean was average of the hourly means.
  millimeter of mercury (mmHg) | 141.1 (7.9) | 140.6 (8.5) | 142.5 (8.8) | 141.6 (7.7) | 143.1 (9.0) | 141.8 (8.4)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline at Month 3 in 24-hour Mean SBP Assessed by ABPM
Description: 24-hour ABPM was programmed to take readings every 20 minutes during the day (6 am to 9:59 pm) and every 30 minutes during the night (10 pm to 5:59 am). An ABPM was considered adequate if: 1. the number of successful daytime readings were ≥33, 2. the number of successful nighttime readings were ≥11, 3. no more than 3 hours are not represented (i.e., 3 sections of 60 minutes where 0 valid readings were obtained). To summarize the 24-hour ABPM, the hourly adjusted mean was calculated. Hourly mean was the average of BP by each hour of the day. The 24-hour mean was the average of the hourly means. Least squares (LS) mean and standard error (SE) were calculated using a mixed model repeated measures (MMRM) approach.
Time Frame: Baseline and Month 3
Population: The Full Analysis Set included all randomized participants who received any amount of the study drug. Overall number analyzed is the number of participants with data available for analyses. As pre-specified in the SAP, for assessment of Month 3 outcome measures, zilebesiran 300mg Q3M and 300mg Q6M were pooled together.
Measure: Least Squares Mean (Standard Error); unit: millimeters of mercury (mmHg)
Groups:
- Zilebesiran 300 mg Q6M and Q3M: Participants received zilebesiran, 300 mg, as SC injection, Q6M or Q3M during the 6-month placebo-controlled DB period. Participants assigned to the Q6M regimen received placebo at Month 3 of the 6-month DB period to maintain the blind. As specified in the SAP, 'Zilebesiran 300 mg Q6M' and 'Zilebesiran 300 mg Q3M' arms were pooled together to report Month 3 analysis.
Arm/Group | Placebo | Zilebesiran 150 mg Q6M | Zilebesiran 300 mg Q6M and Q3M | Zilebesiran 600 mg Q6M
Number analyzed (Participants) | 60 | 68 | 137 | 65
millimeters of mercury (mmHg) | 6.8 (1.58) | -7.3 (1.49) | -10.0 (1.05) | -8.9 (1.52)
Statistical Analysis 1: Comparison: Placebo vs Zilebesiran 300 mg Q6M and Q3M; LS Mean Difference between zilebesiran 300 mg Q6M and placebo, 95% CI was calculated using Dunnett's procedure; Test type: Superiority; p < 0.0001, MMRM — MMRM model included treatment, visit, treatment-by-visit interaction, and race (categorized as Black and all other races) as fixed factors, with baseline 24-hour mean SBP assessed by ABPM as a covariate; Difference in LS Mean = -16.7, 95% CI 2-sided [-21.2 to -12.3], Standard Error of Mean 1.9
Statistical Analysis 2: Comparison: Placebo vs Zilebesiran 600 mg Q6M; The adjusted 95% CI and p-value are based on Dunnett's test. LS Mean Difference between zilebesiran 600 mg Q6M and placebo, 95% CI was calculated using Dunnett's procedure; Test type: Superiority; p < 0.0001, MMRM — The MMRM model included treatment, visit, treatment-by-visit interaction, and race (categorized as Black and all other races) as fixed factors, with baseline 24-hour mean SBP assessed by ABPM as a covariate; Difference in LS Mean = -15.7, 95% CI 2-sided [-20.8 to -10.6], Standard Error of Mean 2.19

2. Secondary Outcome: Change From Baseline at Month 3 in Mean Sitting Office SBP
Description: The mean office BP in the sitting position was used for the analysis. Office BP in the sitting position was collected with a set of 4 replicates. The average of the last 3 replicates was calculated and used for analysis. LS mean and SE were calculated using a MMRM approach.
Time Frame: Baseline and Month 3
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Zilebesiran 150 mg Q6M | Zilebesiran 300 mg Q6M and Q3M | Zilebesiran 600 mg Q6M
Number analyzed (Participants) | 60 | 68 | 133 | 64
mmHg | -0.1 (1.57) | -9.7 (1.49) | -12.1 (1.06) | -9.2 (1.52)
Statistical Analysis 1: Comparison: Placebo vs Zilebesiran 300 mg Q6M and Q3M; Test type: Superiority; p < 0.0001, MMRM — The MMRM model included treatment, visit, treatment-by-visit interaction, and race (categorized as Black and all other races) as fixed factors, with office SBP as a covariate; Tested in hierarchical order with success criterion of nominal p-value <0.05; Difference in LS Mean = -12, 95% CI 2-sided [-15.7 to -8.3], Standard Error of Mean 1.89
Statistical Analysis 2: Comparison: Placebo vs Zilebesiran 600 mg Q6M; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 2, analysis 1]; Tested in hierarchical order with success criterion of nominal p-value <0.05; Difference in LS Mean = -9.1, 95% CI 2-sided [-13.4 to -4.8], Standard Error of Mean 2.19

3. Secondary Outcome: Change From Baseline at Month 6 in 24-hour Mean SBP Assessed by ABPM
Description: 24-hour ABPM was programmed to take readings every 20 minutes during the day (6 am to 9:59 pm) and every 30 minutes during the night (10 pm to 5:59 am). An ABPM was considered adequate if: 1. the number of successful daytime readings were ≥33, 2. the number of successful nighttime readings were ≥11, 3. no more than 3 hours are not represented (i.e., 3 sections of 60 minutes where 0 valid readings were obtained). To summarize the 24-hour ABPM, the hourly adjusted mean was calculated. Hourly mean was the average of blood pressure (BP) by each hour of the day. The 24-hour mean was the average of the hourly means. LS mean and SE were calculated using a MMRM approach.
Time Frame: Baseline and Month 6
Population: The Full Analysis Set included all randomized participants who received any amount of the study drug. Overall number analyzed is the number of participants with data available for analyses.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Zilebesiran 150 mg Q6M | Zilebesiran 300 mg Q6M | Zilebesiran 300 mg Q3M | Zilebesiran 600 mg Q6M
Number analyzed (Participants) | 54 | 62 | 68 | 60 | 63
mmHg | 4.6 (1.73) | -6.5 (1.63) | -9.9 (1.58) | -9.5 (1.65) | -9.6 (1.62)
Statistical Analysis 1: Comparison: Placebo vs Zilebesiran 300 mg Q3M; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 1, analysis 2]; Tested in hierarchical order with success criterion of nominal p-value <0.05; Difference in LS Mean = -14.1, 95% CI 2-sided [-18.9 to -9.4], Standard Error of Mean 2.4
Statistical Analysis 2: Comparison: Placebo vs Zilebesiran 600 mg Q6M; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 1, analysis 2]; Tested in hierarchical order with success criterion of nominal p-value <0.05; Difference in LS Mean = -14.2, 95% CI 2-sided [-18.9 to -9.5], Standard Error of Mean 2.38

4. Secondary Outcome: Change From Baseline at Month 6 in Mean Sitting Office SBP
Description: as for outcome 2
Time Frame: Baseline and Month 6
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Zilebesiran 150 mg Q6M | Zilebesiran 300 mg Q6M | Zilebesiran 300 mg Q3M | Zilebesiran 600 mg Q6M
Number analyzed (Participants) | 57 | 65 | 68 | 57 | 62
mmHg | -0.6 (1.80) | -8.2 (1.70) | -11.1 (1.67) | -12.8 (1.80) | -10.8 (1.73)
Statistical Analysis 1: Comparison: Placebo vs Zilebesiran 300 mg Q3M; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 2, analysis 1]; Tested in hierarchical order with success criterion of nominal p-value <0.05; Difference in LS Mean = -12.1, 95% CI 2-sided [-17.2 to -7.1], Standard Error of Mean 2.55
Statistical Analysis 2: Comparison: Placebo vs Zilebesiran 600 mg Q6M; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 2, analysis 1]; Tested in hierarchical order with success criterion of nominal p-value <0.05; Difference in LS Mean = -10.2, 95% CI 2-sided [-15.1 to -5.3], Standard Error of Mean 2.5

5. Secondary Outcome: Percentage of Participants With 24-hour Mean SBP Assessed by ABPM <130 mmHg and/or Reduction of ≥20 mmHg From Baseline Without Additional Antihypertensive Medications at Month 6
Description: 24-hour ABPM was programmed to take readings every 20 minutes during the day (6 am to 9:59 pm) and every 30 minutes during the night (10 pm to 5:59 am). An ABPM was considered adequate if: 1. the number of successful daytime readings were ≥33, 2. the number of successful nighttime readings were ≥11, 3. no more than 3 hours are not represented (i.e., 3 sections of 60 minutes where 0 valid readings were obtained). To summarize the 24-hour ABPM, the hourly adjusted mean was calculated. Hourly mean was the average of blood pressure (BP) by each hour of the day. The 24-hour mean was the average of the hourly means.
Time Frame: Month 6
Population: The Full Analysis Set included all randomized participants who received any amount of the study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Zilebesiran 150 mg Q6M | Zilebesiran 300 mg Q6M | Zilebesiran 300 mg Q3M | Zilebesiran 600 mg Q6M
Number analyzed (Participants) | 75 | 78 | 73 | 75 | 76
percentage of participants | 6.7 | 30.8 | 50.7 | 38.7 | 47.4
Statistical Analysis 1: Comparison: Placebo vs Zilebesiran 300 mg Q3M; Test type: Superiority; p < 0.0001, Regression, Logistic — Logistic regression model included treatment and race (black; all other races) as factors and baseline 24-hour mean SBP as a covariate; Tested in hierarchical order with success criterion of nominal p-value <0.05; Odds Ratio (OR) = 10.73, 95% CI 2-sided [3.76 to 30.64]
Statistical Analysis 2: Comparison: Placebo vs Zilebesiran 600 mg Q6M; Test type: Superiority; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 5, analysis 1]; Tested in hierarchical order with success criterion of nominal p-value <0.05; Odds Ratio (OR) = 17.93, 95% CI 2-sided [6.24 to 51.52]

6. Secondary Outcome: Change From Baseline at Month 3 in 24-hour Mean DBP Assessed by ABPM
Description: as for outcome 3
Time Frame: Baseline and Month 3
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Zilebesiran 150 mg Q6M | Zilebesiran 300 mg Q6M and Q3M | Zilebesiran 600 mg Q6M
Number analyzed (Participants) | 60 | 68 | 137 | 65
mmHg | 3.5 (0.87) | -4.5 (0.82) | -5.7 (0.58) | -5.8 (0.84)

7. Secondary Outcome: Change From Baseline at Month 6 in 24-hour Mean DBP Assessed by ABPM
Description: 24-hour ABPM was programmed to take readings every 20 minutes during the day (6 am to 9:59 pm) and every 30 minutes during the night (10 pm to 5:59 am). An ABPM was considered adequate if: 1. the number of successful daytime readings were ≥33, 2. the number of successful nighttime readings were≥11, 3. no more than 3 hours are not represented (i.e., 3 sections of 60 minutes where 0 valid readings were obtained). To summarize the 24-hour ABPM, the hourly adjusted mean was calculated. Hourly mean was the average of blood pressure (BP) by each hour of the day. The 24-hour mean was the average of the hourly means. LS mean and SE were calculated using a MMRM approach
Time Frame: Baseline and Month 6
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Zilebesiran 150 mg Q6M | Zilebesiran 300 mg Q6M | Zilebesiran 300 mg Q3M | Zilebesiran 600 mg Q6M
Number analyzed (Participants) | 54 | 62 | 68 | 60 | 63
mmHg | 2.2 (0.97) | -4.8 (0.91) | -6.1 (0.89) | -6.3 (0.93) | -6.3 (0.91)

8. Secondary Outcome: Change From Baseline at Month 3 in Mean Sitting Office DBP
Description: as for outcome 2
Time Frame: Baseline and Month 3
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Zilebesiran 150 mg Q6M | Zilebesiran 300 mg Q6M and Q3M | Zilebesiran 600 mg Q6M
Number analyzed (Participants) | 60 | 68 | 133 | 64
mmHg | -0.6 (1.00) | -5.3 (0.94) | -7.0 (0.67) | -5.4 (0.97)

9. Secondary Outcome: Time Adjusted Change From Baseline Through Month 3 in Mean Sitting Office SBP and DBP
Description: Time adjusted change from baseline in mean sitting office SBP and DBP was the area under the curve (AUC) between Month 1 and 3 visits divided by the duration of time period.
Time Frame: Baseline and Month 3
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Zilebesiran 150 mg Q6M | Zilebesiran 300 mg Q6M and Q3M | Zilebesiran 600 mg Q6M
Number analyzed (Participants) | 60 | 68 | 133 | 64
mmHg
  Office SBP | -0.6 (1.29) | -9.1 (1.24) | -10.9 (0.89) | -10.1 (1.26)
  Office DBP | -0.0 (0.80) | -4.8 (0.77) | -6.5 (0.55) | -6.0 (0.78)

10. Secondary Outcome: Change From Baseline at Month 6 in Mean Sitting Office DBP
Description: as for outcome 2
Time Frame: Baseline and Month 6
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Zilebesiran 150 mg Q6M | Zilebesiran 300 mg Q6M | Zilebesiran 300 mg Q3M | Zilebesiran 600 mg Q6M
Number analyzed (Participants) | 57 | 65 | 68 | 57 | 62
mmHg | -1.2 (1.20) | -4.1 (1.13) | -6.8 (1.12) | -8.2 (1.20) | -5.0 (1.16)

11. Secondary Outcome: Time Adjusted Change From Baseline Through Month 6 in 24-hour Mean SBP and DBP Assessed by ABPM
Description: Time adjusted change from baseline through Month 6 in 24-hour mean SBP and DBP was determined as the AUC between Month 1 and 6 visits divided by the duration of the time period.
Time Frame: Baseline and Month 6
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Zilebesiran 150 mg Q6M | Zilebesiran 300 mg Q6M | Zilebesiran 300 mg Q3M | Zilebesiran 600 mg Q6M
Number analyzed (Participants) | 54 | 62 | 68 | 60 | 63
mmHg
  24-hour Mean SBP | 5.8 (1.26) | -6.3 (1.20) | -9.2 (1.20) | -9.6 (1.22) | -9.1 (1.22)
  24-hour Mean DBP | 3.1 (0.72) | -4.2 (0.69) | -5.5 (0.69) | -5.8 (0.70) | -5.9 (0.70)

12. Secondary Outcome: Time Adjusted Change From Baseline Through Month 6 in Mean Sitting Office SBP and DBP
Description: Time adjusted change is the AUC between Month 1 and 6 visits divided by the duration of time period.
Time Frame: Baseline and Month 6
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Zilebesiran 150 mg Q6M | Zilebesiran 300 mg Q6M | Zilebesiran 300 mg Q3M | Zilebesiran 600 mg Q6M
Number analyzed (Participants) | 57 | 65 | 68 | 57 | 62
mmHg
  Office SBP | -0.5 (1.25) | -9.0 (1.20) | -12.1 (1.21) | -11.0 (1.24) | -10.0 (1.22)
  Office DBP | -0.6 (0.80) | -4.7 (0.76) | -7.2 (0.77) | -6.7 (0.79) | -5.5 (0.78)

13. Secondary Outcome: Change From Baseline in Daytime/Nighttime Mean SBP and DBP Assessed by ABPM at Each Visit
Description: ABPM was programmed to take readings every 20 minutes during the day (6 am to 9:59 pm) and every 30 minutes during the night (10 pm to 5:59 am). An ABPM was considered adequate if: 1. the number of successful daytime readings were ≥33, 2. the number of successful nighttime readings were ≥11, and 3. no more than 3 hours are not represented (i.e., 3 sections of 60 minutes where 0 valid readings were obtained). Baseline was defined as the last assessment prior to receiving the first dose of study drug. LS mean and SE were calculated using a MMRM approach.
Time Frame: Baseline, and Months 1, 3 and 6
Population: The Full Analysis Set included all randomized participants who received any amount of the study drug. Overall number analyzed is the number of participants with data available for analyses. Number analyzed is the number of participants with data available for analyses at specified timepoints.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Zilebesiran 150 mg Q6M | Zilebesiran 300 mg Q6M | Zilebesiran 300 mg Q3M | Zilebesiran 600 mg Q6M
Number analyzed (Participants) | 67 | 72 | 70 | 71 | 69
mmHg
  Change in Daytime Mean SBP at Month 1: number analyzed (Participants) | 67 | 72 | 66 | 71 | 69
  Change in Daytime Mean SBP at Month 1 | 4.3 (1.50) | -3.6 (1.45) | -6.4 (1.51) | -9.6 (1.46) | -9.1 (1.48)
  Change in Daytime Mean SBP at Month 3: number analyzed (Participants) | 60 | 68 | 70 | 67 | 65
  Change in Daytime Mean SBP at Month 3 | 6.7 (1.62) | -7.6 (1.53) | -10.7 (1.52) | -9.8 (1.54) | -8.9 (1.56)
  Change in Daytime Mean SBP at Month 6: number analyzed (Participants) | 54 | 62 | 68 | 60 | 63
  Change in Daytime Mean SBP at Month 6 | 4.5 (1.83) | -6.9 (1.72) | -10.4 (1.66) | -9.3 (1.74) | -8.8 (1.71)
  Change in Nighttime Mean SBP at Month 1: number analyzed (Participants) | 67 | 72 | 66 | 71 | 69
  Change in Nighttime Mean SBP at Month 1 | 4.7 (1.64) | -3.4 (1.59) | -5.1 (1.64) | -9.5 (1.60) | -8.0 (1.62)
  Change in Nighttime Mean SBP at Month 3: number analyzed (Participants) | 60 | 68 | 70 | 67 | 65
  Change in Nighttime Mean SBP at Month 3 | 7.0 (1.85) | -6.4 (1.76) | -8.2 (1.74) | -9.7 (1.77) | -8.5 (1.79)
  Change in Nighttime Mean SBP at Month 6: number analyzed (Participants) | 54 | 62 | 68 | 60 | 63
  Change in Nighttime Mean SBP at Month 6 | 4.7 (1.86) | -5.8 (1.75) | -8.9 (1.69) | -10.2 (1.78) | -11.1 (1.74)
  Change in Daytime Mean DBP at Month 1 | 2.9 (0.91) | -2.7 (0.88) | -4.0 (0.91) | -5.9 (0.89) | -5.8 (0.89)
  Change in Daytime Mean DBP at Month 3: number analyzed (Participants) | 60 | 68 | 70 | 67 | 65
  Change in Daytime Mean DBP at Month 3 | 3.5 (0.94) | -4.8 (0.89) | -6.1 (0.88) | -5.7 (0.90) | -5.6 (0.90)
  Change in Daytime Mean DBP at Month 6: number analyzed (Participants) | 54 | 62 | 68 | 60 | 63
  Change in Daytime Mean DBP at Month 6 | 2.1 (1.07) | -4.8 (1.01) | -6.2 (0.98) | -6.1 (1.02) | -5.7 (1.00)
  Change in Nighttime Mean DBP at Month 1: number analyzed (Participants) | 67 | 72 | 66 | 71 | 69
  Change in Nighttime Mean DBP at Month 1 | 3.2 (1.01) | -2.4 (0.98) | -3.5 (1.02) | -5.9 (0.99) | -5.4 (1.00)
  Change in Nighttime Mean DBP at Month 3: number analyzed (Participants) | 60 | 68 | 70 | 67 | 65
  Change in Nighttime Mean DBP at Month 3 | 3.7 (1.08) | -3.6 (1.02) | -5.1 (1.01) | -4.8 (1.03) | -5.8 (1.04)
  Change in Nighttime Mean DBP at Month 6: number analyzed (Participants) | 54 | 62 | 68 | 60 | 63
  Change in Nighttime Mean DBP at Month 6 | 2.2 (1.09) | -4.3 (1.03) | -5.9 (1.00) | -6.7 (1.05) | -7.6 (1.03)

14. Secondary Outcome: Percentage Change From Baseline in Serum Angiotensinogen (AGT) Through Month 6
Time Frame: Baseline, Week 2 and Months 1, 2, 3, 4, 5 and 6
Population: Pharmacodynamic (PD) Analysis Set included all participants who received at least 1 full dose of study drug. All by-treatment analyses based on the PD Analysis Set were grouped according to the treatment actually received. Overall number analyzed is the number of participants with data available for analyses. Number analyzed is the number of participants with data available for analyses at specified timepoints.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Zilebesiran 150 mg Q6M | Zilebesiran 300 mg Q6M | Zilebesiran 300 mg Q3M | Zilebesiran 600 mg Q6M
Number analyzed (Participants) | 74 | 78 | 73 | 75 | 76
percent change
  Percent Change from Baseline at Week 2: number analyzed (Participants) | 71 | 78 | 72 | 73 | 71
  Percent Change from Baseline at Week 2 | -0.05 (23.99) | -88.34 (9.96) | -92.68 (4.40) | -92.77 (4.03) | -94.49 (5.52)
  Percent Change from Baseline at Month 1: number analyzed (Participants) | 70 | 77 | 73 | 72 | 73
  Percent Change from Baseline at Month 1 | 1.61 (22.96) | -94.48 (9.04) | -97.38 (1.72) | -97.20 (2.30) | -98.22 (2.69)
  Percent Change from Baseline at Month 2: number analyzed (Participants) | 71 | 74 | 72 | 72 | 73
  Percent Change from Baseline at Month 2 | -2.06 (21.87) | -94.47 (12.38) | -97.74 (2.04) | -97.64 (2.15) | -98.70 (0.74)
  Percent Change from Baseline at Month 3: number analyzed (Participants) | 71 | 74 | 72 | 72 | 71
  Percent Change from Baseline at Month 3 | -2.19 (22.86) | -93.31 (9.94) | -97.26 (2.78) | -97.00 (2.61) | -98.25 (1.60)
  Percent Change from Baseline at Month 4: number analyzed (Participants) | 69 | 71 | 71 | 70 | 69
  Percent Change from Baseline at Month 4 | 1.39 (26.06) | -91.89 (11.61) | -95.94 (5.23) | -98.38 (1.08) | -97.98 (1.74)
  Percent Change from Baseline at Month 5: number analyzed (Participants) | 68 | 70 | 70 | 70 | 69
  Percent Change from Baseline at Month 5 | -2.27 (21.18) | -90.10 (12.48) | -94.85 (6.58) | -98.23 (1.13) | -97.38 (2.41)
  Percent Change from Baseline at Month 6: number analyzed (Participants) | 69 | 70 | 70 | 68 | 69
  Percent Change from Baseline at Month 6 | -4.97 (24.90) | -87.84 (13.82) | -93.13 (8.29) | -97.71 (1.91) | -96.41 (4.04)

ADVERSE EVENTS:
Time Frame: 6-Month Placebo-controlled DB Period: Day1 up to Month 6; Post-6-Month DB Period: Pbo/Zil arms: From first zilebesiran dose (Month 6) up to Month 36; Zil/ Zil: From first zilebesiran dose (Day 1) up to Month 36 Placebo-controlled DB: Safety Analysis Set=all participants who received any amount of study drug, grouped per treatment received. As planned, AEs were reported for Zilebesiran Treatment Period using All Zilebesiran Treated Set showing data by treatment sequence (Pbo/Zil & Zil/Zil).
Description: Zilebesiran Treatment Period=Day 1 up to 169 days postdose for zil 150 mg, 300 mg & 600 mg Q6M; up to 85 days postdose for pbo & zil 300 mg Q3M regimes. This Set included all participants receiving any of the 4 zil regimens: those taking zil during 6-month placebo-controlled DB (Zil/Zil) & those switching from pbo to zil after Month 6 (Pbo/Zil). As planned, Zil/Zil arms received same regimen throughout study, so combined AE data are presented for placebo-controlled & Post 6-Month DB periods.
Groups:
- Zilebesiran 300 mg Q6M: Participants received zilebesiran, 300 mg, as SC injection on Day 1 of the 6-month DB period. They received placebo at Month 3 of the 6-month DB period to maintain the blind.
- Zilebesiran/ Zilebesiran 600 mg Q6M: Participants who received zilebesiran 600 mg Q6M during the 6-month placebo-controlled DB period remained on the same regimen throughout the study. Participants received placebo at the visit where no zilebesiran dose was planned to maintain blinding between the Q3M and Q6M regimens.
  Prior to PA6, participants who completed Months 6 to 12 of blinded treatment and pre-dose assessment at Month 12, before a separate OLE study was available, could continue receiving blinded zilebesiran treatment up to additional 24 months in the DB Extension Period. Following PA6, the DB Extension Period was discontinued. Participants who had not yet completed the Month 12 visit at the time of PA6 implementation received their last dose of study drug at Month 9. For participants already in the DB Extension Period at the time of PA6 implementation, dosing depended on scheduled visits: participants whose next visit was at Month 15, 21, 27, or 33 received their planned study drug, while those whose next visit was at Month 18, 24, 30, or 36 did not receive further study drug in the study.
Arm/Group | Placebo | Zilebesiran 150 mg Q6M | Zilebesiran 300 mg Q6M | Zilebesiran 300 mg Q3M | Zilebesiran 600 mg Q6M | Placebo/Zilebesiran 150 mg Q6M | Placebo/Zilebesiran 300 mg Q6M | Placebo/Zilebesiran 300 mg Q3M | Placebo/Zilebesiran 600 mg Q6M | Zilebesiran/Zilebesiran 150 mg Q6M | Zilebesiran/Zilebesiran 300 mg Q6M | Zilebesiran/Zilebesiran 300 mg Q3M | Zilebesiran/ Zilebesiran 600 mg Q6M
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/78 | 0/73 | 1/75 | 0/76 | 0/16 | 0/16 | 0/16 | 0/18 | 1/78 | 0/73 | 1/75 | 0/76
Serious Adverse Events (participants affected / at risk) | 5/75 | 0/78 | 1/73 | 4/75 | 6/76 | 1/16 | 0/16 | 1/16 | 0/18 | 5/78 | 5/73 | 7/75 | 9/76
Other Adverse Events (participants affected / at risk) | 18/75 | 21/78 | 24/73 | 23/75 | 20/76 | 9/16 | 12/16 | 9/16 | 8/18 | 53/78 | 47/73 | 49/75 | 49/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=75) | Zilebesiran 150 mg Q6M (N=78) | Zilebesiran 300 mg Q6M (N=73) | Zilebesiran 300 mg Q3M (N=75) | Zilebesiran 600 mg Q6M (N=76) | Placebo/Zilebesiran 150 mg Q6M (N=16) | Placebo/Zilebesiran 300 mg Q6M (N=16) | Placebo/Zilebesiran 300 mg Q3M (N=16) | Placebo/Zilebesiran 600 mg Q6M (N=18) | Zilebesiran/Zilebesiran 150 mg Q6M (N=78) | Zilebesiran/Zilebesiran 300 mg Q6M (N=73) | Zilebesiran/Zilebesiran 300 mg Q3M (N=75) | Zilebesiran/ Zilebesiran 600 mg Q6M (N=76)
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Obstructive pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Endocarditis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Coronary bypass stenosis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Breast cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Malignant melanoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Paraganglion neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abnormal behaviour (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aortic aneurysm (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertensive urgency (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=75) | Zilebesiran 150 mg Q6M (N=78) | Zilebesiran 300 mg Q6M (N=73) | Zilebesiran 300 mg Q3M (N=75) | Zilebesiran 600 mg Q6M (N=76) | Placebo/Zilebesiran 150 mg Q6M (N=16) | Placebo/Zilebesiran 300 mg Q6M (N=16) | Placebo/Zilebesiran 300 mg Q3M (N=16) | Placebo/Zilebesiran 600 mg Q6M (N=18) | Zilebesiran/Zilebesiran 150 mg Q6M (N=78) | Zilebesiran/Zilebesiran 300 mg Q6M (N=73) | Zilebesiran/Zilebesiran 300 mg Q3M (N=75) | Zilebesiran/ Zilebesiran 600 mg Q6M (N=76)
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thyroid mass (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Glaucoma (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 2 | 3 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 3 | 2 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 3 | 0 | 2
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 2
Discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 2 | 3
Injection site reaction (General disorders) | 0 | 3 | 4 | 8 | 4 | 0 | 3 | 1 | 1 | 5 | 8 | 13 | 9
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 2 | 1 | 2
Coronavirus Disease of 2019 (COVID-19) (Infections and infestations) | 3 | 3 | 6 | 6 | 4 | 0 | 1 | 0 | 0 | 7 | 7 | 9 | 8
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 5 | 2
Onychomycosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia mycoplasmal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 4 | 3
Upper respiratory tract infection (Infections and infestations) | 1 | 3 | 4 | 2 | 1 | 2 | 0 | 1 | 1 | 6 | 5 | 6 | 4
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 1 | 3 | 5 | 9 | 3
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Brain contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 1 | 0 | 0
Muscle injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood creatine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 2 | 0 | 1
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1
Glomerular filtration rate decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1
Glycosylated haemoglobin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 2 | 3
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 5 | 4 | 5 | 5 | 0 | 1 | 0 | 0 | 6 | 5 | 7 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 4 | 2 | 0 | 0 | 0 | 0 | 2 | 3 | 6 | 4 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 3 | 3 | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 3 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 3 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 3 | 1
Dizziness (Nervous system disorders) | 4 | 2 | 2 | 3 | 3 | 0 | 0 | 0 | 1 | 3 | 3 | 4 | 8
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 7 | 0 | 4 | 2 | 1 | 0 | 0 | 0 | 0 | 2 | 6 | 5 | 3
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Renal cyst (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 1
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 5 | 4 | 0 | 3 | 5 | 1 | 0 | 1 | 0 | 9 | 3 | 4 | 9
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 1 | 2 | 2
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2024-09-06): https://cdn.clinicaltrials.gov/large-docs/35/NCT04936035/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-05): https://cdn.clinicaltrials.gov/large-docs/35/NCT04936035/SAP_001.pdf